CLINICAL TRIAL: NCT02786823
Title: Effect of Folic Acid and Vitamin B12 Supplementation on Biochemical Parameters in Subjects With Type-2 Diabetes
Brief Title: Effect of Folic Acid and Vitamin B12 Supplementation in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Debapriya Bandyopadhyay, Assistant Professor, Department of Biochemistry, All India Institute of Medical Sciences, Bhubaneswar, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: T/lM-F/Biochem/15/22
Record Dates: First submitted 2016-05-25; First posted 2016-06-01 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Folic Acid; Vitamin B 12; Hypoglycemic Agents; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Folic acid (Experimental): Twenty type-2 diabetes patients with standard Oral hypoglycemic agents [Metformin +/- Sulfonylurea] will be recruited and additionally receive tab. Folic acid 5 mg once daily for 8 weeks
  Interventions: Dietary Supplement: Folic acid; Drug: Oral hypoglycemic agents [Metformin +/- Sulfonylurea]
- Vitamin B12 (Experimental): Twenty type-2 diabetes patients with standard Oral hypoglycemic agents [Metformin +/- Sulfonylurea] will be recruited and additionally receive tab. Vitamin B12 500 mcg once daily for 8 weeks
  Interventions: Dietary Supplement: Vitamin B12; Drug: Oral hypoglycemic agents [Metformin +/- Sulfonylurea]
- "Folic acid" and "Vitamin B12" (Experimental): Twenty type-2 diabetes patients with standard Oral hypoglycemic agents [Metformin +/- Sulfonylurea] will be recruited and additionally receive both tab. Folic acid 5 mg once daily and tab. Vitamin B12 500 mcg once daily for 8 weeks
  Interventions: Dietary Supplement: Folic acid; Dietary Supplement: Vitamin B12; Drug: Oral hypoglycemic agents [Metformin +/- Sulfonylurea]
- Control (Active Comparator): Twenty type-2 diabetes patients with standard Oral hypoglycemic agents [Metformin +/- Sulfonylurea] will be recruited and receive no additional supplementation
  Interventions: Drug: Oral hypoglycemic agents [Metformin +/- Sulfonylurea]

INTERVENTIONS:
Dietary Supplement: Folic acid — tab. Folic acid 5 mg
  Arms: "Folic acid" and "Vitamin B12"; Folic acid
Dietary Supplement: Vitamin B12 — tab. Vitamin B12 500 mcg
  Arms: "Folic acid" and "Vitamin B12"; Vitamin B12
Drug: Oral hypoglycemic agents [Metformin +/- Sulfonylurea] — Patients receiving either of the following oral hypoglycemic agents
  1. Sulfonylurea
  2. Metformin
  3. Metformin plus Sulfonylurea
  Other Names: Metformin, Sulfonylurea

SUMMARY:
This study aims to evaluate the effect of Folic acid and Vitamin B12 supplementation on Biochemical parameters in subjects with type-2 Diabetes. 80 selected subjects will be divided into 4 groups of 20 each.

* Group A: to receive Folic acid 5 mg once daily for 8 weeks along with standard oral anti-diabetic drugs;
* Group B: to receive Vitamin B12 500 mcg once daily for 8 weeks along with standard oral anti-diabetic drugs;
* Group C: to receive both Folic acid 5 mg once daily and Vitamin B12 500 mcg once daily for 8 weeks along with standard oral anti-diabetic drugs;
* Group D: to receive no additional intervention apart from standard oral anti-diabetic drugs.

The biochemical parameters will be evaluated before and after the intervention.

DETAILED DESCRIPTION:
This is a randomized, parallel group, open label study to evaluate the effect of Folic acid and Vitamin B12 supplementation on Biochemical parameters in subjects with type-2 Diabetes.

80 selected subjects will be randomly assigned to 4 groups of 20 each as follows:

* Group A: to receive Folic acid 5 mg once daily for 8 weeks along with standard oral anti-diabetic drugs;
* Group B: to receive Vitamin B12 500 mcg once daily for 8 weeks along with standard oral anti-diabetic drugs;
* Group C: to receive both Folic acid 5 mg once daily and Vitamin B12 500 mcg once daily for 8 weeks along with standard oral anti-diabetic drugs;
* Group D: to receive no additional intervention apart from standard oral anti-diabetic drugs.

The subjects will also be advised to be on a normal routine diet, not to skip any meal and not to change their exercise pattern (if any) during the study period.The compliance of the intervention will be monitored by instructing the patients to return all unused tablets at the end of the 8 weeks period of study.

All the subjects will be asked to report after an overnight fasting of 12 hours on two occasions i.e. at the start of the study before allocation of group and 8 weeks after allocation. After measurement of body weight, height and blood pressure (by Mercury Sphygmomanometer), 5 milliliter of early morning fasting venous blood sample will be collected under aseptic measures on both the occasions. The samples collected will then be appropriately processed for the analysis of various biochemical parameters.

The results of all the parameters evaluated will be recorded in the subject's Data Collection Form.The data will be analyzed using Statistical Package for the Social Sciences (SPSS) version 21.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetic patients within age group 30-65 years, on stable dose of anti-diabetic with/without anti-hypertensive drugs will be included in this study

Exclusion Criteria:

* Subjects on non-allopathic forms of treatment for diabetic control.
* Subjects with Chronic Renal disease and Liver disease.
* Subjects with malabsorption.
* Subjects with Thyroid function abnormalities.
* HbA1c levels more than 10 %
* Smoking
* Alcoholism
* Pregnant subjects
* Subjects with vitamin B12 deficiency
* Subjects already on Folate or Vitamin B12 supplementation due to some other medical condition
* The detailed drug history of the subjects will be taken prior to including them in the study. Antibiotics like Fluoroquinolones; anti-seizure drugs like phenytoin; Corticosteroids and Hormonal Contraceptives; Hypolipidemic drugs like statins are known to affect Glucose metabolism and subjects on these medications will not be included in the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
HbA1c | 8 weeks

SECONDARY OUTCOMES:
Fasting plasma glucose | 8 weeks
Fasting plasma insulin | 8 weeks
Insulin Resistance | 8 weeks
  Using Homeostatic model assessment (HOMA2 calculator which uses fasting plasma glucose and plasma insulin values to calculate insulin resistance)
Serum total cholesterol | 8 weeks
Serum triacylglycerol | 8 weeks
Serum Low-density lipoprotein (LDL) | 8 weeks
Serum High-density lipoprotein (HDL) | 8 weeks
Serum Very Low-density lipoprotein (VLDL) | 8 weeks
Serum Homocysteine | 8 weeks
Serum Adiponectin | 8 weeks
Serum Tumor Necrosis Factor (TNF) | 8 weeks
Serum Interleukin-6 (IL-6) | 8 weeks
Serum C reactive protein (CRP) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Debapriya Bandyopadhyay, M.D., Principal Investigator — All India Institute of Medical Sciences, Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Bhubaneswar, Odisha, India